CLINICAL TRIAL: NCT05407246
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase II Clinical Study on the Efficacy and Safety of hemay005 Tablets in the Treatment of Active Ankylosing Spondylitis
Brief Title: Phase II Study of Hemay005 in Patients With Active Ankylosing Spondylitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Hemay Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Organization: Ganzhou Hemay Pharmaceutical Co., Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HM005AS2S01
Record Dates: First submitted 2022-05-30; First posted 2022-06-07 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Active Ankylosing Spondylitis
MeSH Terms: interventions — Hemay005

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hemay005 75mg BID group (Active Comparator): 75mg BID of Hemay005; daily oral administrtion for 16 weeks
  Interventions: Drug: Hemay005
- Hemay005 60mg BID group (Active Comparator): 60mg BID of Hemay005; daily oral administrtion for 16 weeks
  Interventions: Drug: Hemay005
- placebo group (Placebo Comparator): Placebo of Hemay005; daily oral administrtion for 16 weeks
  Interventions: Drug: Hemay005

INTERVENTIONS:
Drug: Hemay005 — Hemay005 60 mg treatment group (group A): hemay005 tablets 60 mg bid were used during the treatment period; Hemay005 75 mg treatment group (group B): hemay005 75 mg bid was used during the treatment period; Placebo group (Group C): placebo (hemay005 tablet simulant) bid was used during the treatment period;
  Other Names: placebo

SUMMARY:
This study is a multicenter, randomized, double-blind, placebo-controlled phase II clinical study. The study was divided into three stages, including screening period(4-week), treatment period(16-week) and observation period. All subjects need to enter a 28 day (4-week) observation period after stopping hemay005 treatment.

Main purpose:

The efficacy of hemay005 tablet in the treatment of active ankylosing spondylitis (as) was evaluated by placebo parallel control.

Secondary purpose:

* To evaluate the safety of oral hemay005 tablets in patients with active as.
* To evaluate the population pharmacokinetics of hemay005 tablets in patients with active as.

DETAILED DESCRIPTION:
This study is a multicenter, randomized, double-blind, placebo-controlled phase II clinical study. The study was divided into three stages, including screening period, treatment period and observation period. All subjects need to enter a 28 day (4-week) observation period after stopping hemay005 treatment.

Screening period: all subjects shall have a screening period of no more than 28 days (4 weeks) before the baseline visit (day 1 of randomization).

Treatment period: after screening and meeting the inclusion requirements of the study, as subjects were randomly divided into hemay005 60 mg twice daily (bid) dose group (group A), 75 mg bid dose group (group B) and placebo control group (Group C) according to the ratio of 1:1:1. A total of 90 subjects were included in the three groups. They were titrated in the first 6 days. From the 7th day, the subjects received fixed dose administration twice a day for 112 consecutive days (16 weeks). Considering the difference in the proportion of men and women with as, and the slow onset and mild condition of women, randomization will minimize the imbalance between treatment groups according to gender stratification.

Observation period: Subjects in the study (including those who withdrew from the treatment early for any reason) shall be observed for 4 weeks after the end of the last administration.

Main purpose:

The efficacy of hemay005 tablet in the treatment of active ankylosing spondylitis (as) was evaluated by placebo parallel control.

Secondary purpose:

* To evaluate the safety of oral hemay005 tablets in patients with active as.
* To evaluate the population pharmacokinetics of hemay005 tablets in patients with active as.

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign the informed consent form of this study.
* Aged between 18 and 65 years old (both ends included, subject to the date of signing the informed consent form), male or female.
* 50 kg ≤ male weight <100 kg, 45 kg ≤ female weight <100 kg.
* The results of human leucocyte antigen (HLA) -b27 were positive.
* Be able to comply with the follow-up schedule and other protocol requirements
* As (revised New York standard 1984) was diagnosed as follows:

  1. Low back pain lasted for at least 3 months. The pain improved with activity, but the rest did not reduce;
  2. The movement of lumbar vertebra in the direction of anteroposterior and lateral flexion was limited;
  3. The extension range of thorax was smaller than the normal value of the same age and sex;
  4. Bilateral sacroiliac arthritis grade II ~ IV, or unilateral sacroiliac arthritis grade III ~ IV.

If the patient has 4) and adds any one of 1) ~3) respectively, it can be diagnosed as as;

* The subjects shall at least meet the requirements of 1) and 2) below:

  1. Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) ≥ 4, and chronic low back pain ≥ 4 (patient back pain intensity assessment question 1) (NRS score);
  2. At least one nonsteroidal anti-inflammatory drugs (NSAIDs) was used before randomization, but the symptoms were not relieved or the drugs were intolerable or there were drug contraindications, that is, at least 4 weeks of stable use of 1 NSAID at the recommended dose or ≥ 2 NSAIDs, each NSAID was used stably for ≥ 2 weeks) or intolerable before randomization;
  3. In case of any of the following three criteria, the subject shall also meet the corresponding provisions:

  <!-- -->

  1. Patients who are receiving NSAIDs, oral glucocorticoids (prednisone with daily oral glucocorticoid dose ≤ 10 mg or other equivalent dose) and / or cyclooxygenase-2 (COX-2) inhibitors, the dosage is stable at least 14 days before randomization and throughout the study period;
  2. For patients with combined use of sulfasalazine: subjects who began to take sulfasalazine [≤ 3 g/ day] at least 12 weeks before randomization and whose dose and route of administration have been stable for at least 4 weeks before randomization can continue to take sulfasalazine at a sustained dose during the study period;
  3. For previous use of tumor necrosis factor (TNF)- α Patients with inhibitors: TNF α Subjects with inhibitors did not respond adequately to the approved dose for at least 12 weeks, or did not tolerate the treatment;
* The following laboratory standards must be met:

Hemoglobin (HB) ≥ 9 g/dl Hematocrit ≥ 27% White blood cell (WBC) count ≥ 3000/ μ L（≥3.0 × 109/l) and <20000/ μ L（<20 × 109/L） Neutrophil (neu) ≥ 1500/ μ L（≥1.5 × 109/L） Platelet (PLT) ≥ 100000/ μ L（≥100 × 109/L） Serum creatinine (CR) ≤ 1.5 mg/dl (≤ 132.6 μ mol/L) Total bilirubin (TBIL) ≤ 2.0 mg/dl Aspartate aminotransferase, AST (serum glutamic oxaloacetic transaminase, SGOT) and alanine aminotransferase, ALT (serum glutamic pyruvic transaminase, SGPT)] ≤ 1.5 times the upper limits of normal (ULN);

• During the whole study period since the signing of the informed consent and within 3 months after the last administration of the study drug, Female subjects with fertility and male subjects without vasectomy are willing to take effective contraceptive measures [effective contraceptive measures include vasectomy, abstinence, intrauterine device (IUD), hormones (oral, patch, ring, injection, implantation) and barrier method (diaphragm, cervical cap, sponge, condom)]; The serum pregnancy test [human chorionic gonadotropin (hCG)] of fertile female subjects within the first 7 days of randomization must be negative; Male subjects could not donate sperm within 3 months after the first administration of the study drug to the last Administration [Note: fertility is defined as: non menopausal women who have experienced menarche, have not undergone sterilization (hysterectomy / bilateral oophorectomy / bilateral tubal ligation), and have undergone sterilization but have not completed 6 months (menopause refers to continuous natural menopause ≥ 12 months)].

Exclusion Criteria:

* Have the following diseases or disease history:

  1. Complete rigidity of spine or complete fusion of sacroiliac joint;
  2. Patients with a history of other rheumatic autoimmune diseases (such as systemic lupus erythematosus, rheumatoid arthritis, etc.);
  3. Patients with a history of tuberculosis or active tuberculosis (there are signs or symptoms of active tuberculosis judged by the researcher at the time of screening):

     If the patient has a previous history of tuberculosis and has been cured for at least 3 years before randomization according to the researcher's assessment, screening is allowed; Subjects with negative T-SPOT during screening can be included in this study. Subjects with positive T-SPOT in the screening period need to undergo tuberculosis related clinical examination (tuberculosis related clinical examination conducted within 12 weeks before randomization can be directly used for evaluation). If tuberculosis related clinical examination is confirmed as active tuberculosis, subjects cannot be selected for this study; If tuberculosis related clinical examination confirms inactive tuberculosis, the subject can be included in this study. If the research center is unable to carry out T-SPOT test, it can also accept tuberculosis screening with QuantiFERON TB gold test kit. The processing of QuantiFERON TB gold screening results is the same as that of T-SPOT;
  4. Patients with malignant tumor or any history of malignant tumor within 5 years before screening (except skin squamous cell carcinoma in situ, basal cell carcinoma or cervical carcinoma in situ after treatment and no recurrence evidence in the past 12 weeks);
  5. Evidence of active infection within 1 month before screening, including acute and chronic infection and local infection, such as sepsis, abscess, cellulitis and opportunistic fungal (such as Candida) infection (which can be judged by the research doctor in combination with the specific situation of the patient);
  6. Patients with severe basic diseases, such as heart, lung, kidney, liver, nerve, endocrine, gastrointestinal, metabolic or hematological diseases, moderate to severe congestive heart failure (New York Heart Association grade III or IV);
  7. Have a history of alcohol or drug abuse or dependence, or a history of mental illness;
  8. Situations that may affect the absorption of oral drugs, such as subtotal gastrectomy, clinically significant diabetes gastroenteropathy, or some types of weight loss surgery such as gastric bypass surgery, do not include operations that simply partition the stomach into a separate chamber, such as gastric banding surgery;
* Pregnant or lactating women;
* Those who are allergic or allergic to the study drug or its preparation components;
* Those who have undergone major surgery (including spinal surgery or joint surgery) within the first 6 months or plan to undergo major surgery during the trial;
* Those who have participated in clinical trials of any drugs or medical devices within the first three months of screening;
* Those who plan to receive attenuated or live vaccine during the test;
* Taking or having the following medication history:

  1. Patients who used disease modifying anti rheumatic drugs (DMARDs) methotrexate, penicillamine, sulfasalazine, azathioprine and hydroxychloroquine within the first 4 weeks of randomization, except those who used sulfasalazine at a stable dose, and other unlisted abiotic agents were eluted according to 5 drug half lives (or 4 weeks, whichever is longer);
  2. Intravenous or articular endothelium steroids were used within the first 4 weeks of randomization;
  3. Etanercept, adalimumab, efuzumab, infliximab and afacept were used within 8 weeks before randomization, and other unlisted biological agents were eluted according to 5 drug half lives (or 8 weeks, whichever is longer);
  4. Those who used apster before randomization;
  5. Those who used strong cytochrome P450 enzyme inducers within 4 weeks before randomization (e.g., rifampicin, phenobarbital, carbamazepine, phenytoin sodium);
  6. Those who used Tripterygium Wilfordii and other proprietary Chinese medicine or traditional Chinese medicine decoction within 2 weeks before randomization;
* There are any clinically significant abnormalities in 12 lead ECG at the time of screening, and the researcher assessed that participating in this study may increase the risk of subjects or interfere with data interpretation;
* Patients with clinically significant abnormalities in chest X-ray (CXR) or computed tomography (CT) during screening, and the researchers may put the subjects at safety risk;
* subjects with positive hepatitis B B surface antigen (HBsAg), hepatitis C virus antibody (HCVAb), human immunodeficiency virus antibody (hivab) or Treponema pallidum antibody;
* Have committed suicide (including active attempt, interrupted attempt or attempted attempt) or have suicidal thoughts in the past 6 months;
* The researcher believes that there are any other circumstances that are not suitable for participating in the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-08-05 (Actual); Primary Completion 2023-08-18 (Actual); Study Completion 2023-08-18 (Actual)

PRIMARY OUTCOMES:
ASAS20 | week 16
  The proportion of subjects who achieved ASAS 20 remission at the week 16，higher proportion means better effecacy of Hemay005.

SECONDARY OUTCOMES:
BASFI | week 2, 4, 8, 12 and 16
  Changes of Ankylosing Spondylitis Functional Index (BASFI), the more scores change means a better outcome.
BASDAI | week 2, 4, 8, 12 and 16
  Changes of Ankylosing Spondylitis Functional Index (BASDAI),the more scores change means a better outcome.
ASAS20 | week 2, 4, 8, 12
  The proportion of subjects who achieved ASAS 20 remission,higher proportion means better effecacy of Hemay005.
ASAS40 | week 2, 4, 8, 12 and 16
  The proportion of subjects who achieved ASAS 40 remission,higher proportion means better effecacy of Hemay005.
ASQoL | week 16
  Changes in total scores of ankylosing spondylitis quality of life (asqol),the more scores change means a better outcome.
BASMI | week 2, 4, 8, 12 and 16
  Changes in the Bath Ankylosing Spondylitis measurement index (BASMI),the more scores change mean a better outcome.
hs-CPR | week 2, 4, 8, 12 and 16
  Changes of hypersensitive C-reactive protein (hs CRP) ;
MASES | week 2, 4, 8, 12 and 16
  Changes of Maastricht ankylosing spondylitis adhesion score (MASES),the more scores change mean a better outcome.
Extraarticular manifestations | week 2, 4, 8, 12 and 16
  Extraarticular manifestations,,(Such as uveitis, inflammatory bowel disease and psoriasis), and record the history (existence) of these manifestations and the new occurrence or deterioration of these manifestations;
ESR | week 2, 4, 8, 12 and 16
  Changes of erythrocyte sedimentation rate (ESR) in acute phase;

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofeng Zeng, M.D, Principal Investigator — Peking Union Medical College
Locations (11):
- China (11):
  - The First Affiliated Hospital of Bengbu Medical University, Hefei, Anhui
  - Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - The Third Affiliated Hospital of Sun Yat sen University, Guangzhou, Guangdong
  - Hebei CNPC Central Hospital, Langfang, Hebei
  - Puyang Oilfield General Hospital, Puyang, Henan
  - Tongji Hospital Affiliated to Tongji Medical College of Huazhong University of science and technology, Wuhan, Hubei
  - Chenzhou first people's Hospital, Chenzhou, Hunan
  - Pingxiang people's Hospital, Pingxiang, Jiangxi
  - Jilin Provincial People's Hospital, Changchun, Jilin
  - The First Affiliated Hospital of Medical College of Xi'an Jiaotong University, Xi’an, Shanxi

IPD SHARING:
Plan to Share IPD: No
It is yet decided not to share the individual participant data (IPD) to other researchers.